CLINICAL TRIAL: NCT01215422
Title: Anesthesiologists Learning to Use Videolaryngoscopes in Children
Brief Title: Success of Pediatric Anesthesiologists in Learning to Use Videolaryngoscopes
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: Verathon (Industry); KARL STORZ Endoscopy-America, Inc. (Industry)
Responsible Party: Principal Investigator, Joan Robinson, Physician, University of Alberta
Other Study IDs: JR-01
Record Dates: First submitted 2010-10-04; First posted 2010-10-06 (Estimated); Results first posted 2012-10-08 (Estimated); Last update posted 2012-10-08 (Estimated); Status verified 2012-10

CONDITIONS: Tracheal Intubation Morbidity
Keywords: Surgical procedures; Intubation; Anesthesiologist; Laryngoscope; Videolaryngoscope

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- children intubated with Glidescope: children intubated with Glidescope
  Interventions: Procedure: timed intubation
- children intubated with DCI: children intubated with DCI
  Interventions: Procedure: timed intubation

INTERVENTIONS:
Procedure: timed intubation — timed intubation

SUMMARY:
There are two new instruments on the market that anesthesiologists use when putting a breathing tube into the lungs of patients. The purpose of this study is to see how easily anesthesiologists can learn to use them in children.

DETAILED DESCRIPTION:
Each anesthesiologist performed 20 timed baseline intubations. They were then randomized to perform 20 timed intubations with one of the two new videolaryngoscopes followed by 20 with the other new videolaryngoscope. The goal was to see how quickly they could become proficient.

ELIGIBILITY:
Inclusion Criteria for Children Population:

- Children requiring intubation for elective or non-elective surgery

Exclusion Criteria:

* Children with raised intracranial pressure
* Children with potential cervical spine injuries
* Children at risk for regurgitation because of a full stomach
* Children who were anticipated to have a difficult airway based on their physical appearance or previous experience were excluded.

Inclusion Criteria for Anesthesiologist Population:

*Anesthesiologists who care for children at Stollery Children's Hospital

Exclusion Criteria for Anesthesiologist Population:

*None

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children being intubated for surgery
Sampling Method: Non-Probability Sample
Enrollment: 646 (Actual)
Dates: Start 2007-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan L Robinson, MD, Principal Investigator — University of Alberta
Locations (1):
- Stollery Children's Hospital, Edmonton, Alberta, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children were recruited pre-op if their anesthesiologist was participating in the study. Anesthesiologists did 20 baseline intubations with a standard laryngoscope and then were randomized to use the GlideScope(GS)or Karl Storz Direct Coupled Interface (KS) video laryngoscope (VLS) for 20 intubations), followed by the other VLS.
Pre-assignment Details: Patients with anticipated difficult airways were excluded.
Groups:
- Overall Anesthesiologists: Baseline intubation times were obtained on a convenience sample of 20 children using the standard laryngoscope blade of their choice. Then anesthesiologists were randomized to complete either 20 intubations with the GlideScope system (GS) video laryngoscope (VLS) or 20 with the Karl Storz Direct Coupled Interface DCI (KS) VLS first. Once they had intubated 20 children with the VLS to which they were randomized, they crossed over to use the alternate VLS for 20 intubations.
- Baseline Intubation Participants: Children intubated at baseline using the standard laryngoscope blade of the anesthesiologist's choice.
- KS Intubation Participants: Children intubated with the Karl Storz Direct Coupled Interface DCI (KS) VLS
- GS Intubation Participants: Children intubated with the GlideScope system (GS) VLS
Period: Overall Study
Arm/Group | Overall Anesthesiologists | Baseline Intubation Participants | KS Intubation Participants | GS Intubation Participants
Started | 14 | 249 | 196 | 201
Completed | 6 | 249 | 193 | 193
Not Completed | 8 | 0 | 3 | 8
Not completed — Relocation | 1 | 0 | 0 | 0
Not completed — Failed intubations | 0 | 0 | 3 | 8
Not completed — Did not complete all intubations | 7 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- KS Intubation Participants: Children intubated with the Karl Storz Direct Coupled Interface (DCI) (KS) video laryngoscope (VLS)
- GS Intubaton Participants: Children intubated with the GlideScope system (GS) video laryngoscope (VLS)
- Total: Total of all reporting groups
Arm/Group | Overall Anesthesiologists | Baseline Intubation Participants | KS Intubation Participants | GS Intubaton Participants | Total
Number analyzed (Participants) | 13 | 249 | 196 | 201 | 659
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 249 | 196 | 201 | 646
  Between 18 and 65 years | 13 | 0 | 0 | 0 | 13
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: participants] — Gender of the children was not recorded as it was not thought to be of relevance for intubation participants.
  participants
    Unknown | 0 | 249 | 196 | 201 | 646
    Male | 6 | 0 | 0 | 0 | 6
    Female | 7 | 0 | 0 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Success in Learning to Use a Videolaryngoscope(VLS)
Description: Anesthesiologists were to perform 20 intubations with each videolaryngoscopes. #1-10 were for practice. "Rapid Success" was no failed intubation attempts on #11-20 and a median time-to-intubation no more than 50% longer than their baseline median time-to-intubation on #11-15 . "Delayed Success" was achieving these same parameters on #16-20 if they were not achieved on #11-15. Operators who did not achieve either goal were labeled as having "No Success".
Time Frame: Up to 5 minutes per intubation
Population: Only anesthesiologists who completed minimum 18 intubations with either laryngoscope were analyzed for the primary outcome.
Measure: Number; unit: percent of anesthesiologists
Units Other Than Participants: intubations
Groups:
- GS Intubations: Anesthesiologists who performed minimum 18 intubations with the GS VLS.
- KS Intubations: Anesthesiologists who performed minimum 18 intubations with the KS VLS
Arm/Group | GS Intubations | KS Intubations
Number analyzed (Participants) | 8 | 8
Number analyzed (intubations) | 193 | 193
percent of anesthesiologists
  Rapid Success | 37.5 | 62.5
  Delayed Success | 25 | 0
  No Success | 37.5 | 37.5
Statistical Analysis 1: Comparison: GS Intubations vs KS Intubations; Test type: Superiority or Other; p > 0.05, Regression, Logistic; Odds Ratio (OR) = 2, 95% CI 1-sided [lower limit 0.15]

2. Secondary Outcome: Cormack & Lehane Score
Description: This Outcome was designed to determine if the view of the airway as determined by the Cormack & Lehane grading system is improved by use of the GlideScope (GS) video laryngoscope and/or the Karl Storz Direct Coupled Interface (DCI) (KS) video laryngoscope as this would be a surrogate marker for utility in a difficult airway. Score is reported as a whole number from I to IV with I being an easy intubation and IV being one where the larynx cannot be visualized at all.
Time Frame: reported during intubation (up to 5 minutes)
Population: Patients were excluded if the Cormack-Lehane score was not recorded.
Measure: Number; unit: Percentage of participants
Groups:
- GS Intubation Participants: Children intubated with the GlideScope system (GS) video laryngoscope (VLS)
- Baseline Intubation Participants: Children intubated at baseline using the standard laryngoscope of the anesthesiologist's choice
Arm/Group | GS Intubation Participants | KS Intubation Participants | Baseline Intubation Participants
Number analyzed (Participants) | 199 | 194 | 249
Percentage of participants
  Grade I | 80.3 (0.46) | 82.5 (0.44) | 84.3 (0.49)
  Grade II | 19.7 | 16.5 | 12.0
  Grade III | 0 | 0.5 | 3.2
  Grade IV | 0 | 0 | 0.4
Statistical Analysis 1: Comparison: GS Intubation Participants vs KS Intubation Participants vs Baseline Intubation Participants; Test type: Superiority or Other; p = 0.03, Fisher Exact — The p-value represents the comparison of the two interventions combined and compared against baseline for Grades III and IV summed together

3. Secondary Outcome: Time to Intubation, Analyzed by Order of Laryngoscopes Used
Description: To determine if the learning curve was altered by the order in which the two new laryngoscopes were learned by the anesthesiologist,mean and median times on intubations #16-20 were compared for the two videolaryngoscopes.
Time Frame: 4 years
Population: Only anesthesiologists who completed minimum 18 intubations with each scope were included. We report the mean of their mean times and the mean of their median times on intubations #16-20 when they should have attained a reasonable skill level.
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: anesthesiologists
Arm/Group | GS Intubation Times for Those Who Used GS First | KS Intubation Times for Those Who Used KS First | GS Intubation Times for Those Who Used KS First | KS Intubation Times for Those Who Used GS First
Number analyzed (Participants) | 3 | 3 | 3 | 3
Number analyzed (anesthesiologists) | 3 | 3 | 3 | 3
seconds
  Average of median times | 31.0 (4.8) | 22.2 (1.6) | 25.6 (1.0) | 27.5 (4.2)
  Average of mean times | 30.7 (4.5) | 23.7 (2.4) | 27.4 (2.3) | 30.8 (5.2)

4. Secondary Outcome: Time to Intubation, Stratified by Weight of Patients
Description: To compare the time-to-intubation for these laryngoscopes in children of different weights.
Time Frame: 4 years
Population: Time to Intubation, Stratified by Weight of Patients
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- GS Intubation Participants: Children successfully intubated with the GlideScope system (GS) video laryngoscope (VLS)
- KS Intubation Participants: Children successfully intubated with the Karl Storz Direct Coupled Interface (DCI) (KS) video laryngoscope (VLS)
- Baseline Intubation Participants: Children intubated with the standard laryngoscope of the anesthesiologist's choice
Arm/Group | GS Intubation Participants | KS Intubation Participants | Baseline Intubation Participants
Number analyzed (Participants) | 193 | 193 | 249
seconds
  < 10 kg Body Weight (n=12,9,32) | 33.9 (12.1) | 26.9 (8.4) | 23.8 (7.8)
  >=10 kg Body Weight (n=181,184,217) | 30.0 (10.8) | 28.8 (10.5) | 20.2 (9.4)

5. Secondary Outcome: Mean Years Since Completion of Anesthesiology Residency
Description: To investigate whether there was a correlation between the years since completion of anesthesiology residency to the mid-point of study (2008)and median time-to-intubation for all first attempt intubations for the study. Years since completion of anesthesiology residency reported in the data table, correlation reported in the statistical analysis below
Time Frame: Baseline (assessed as of 2008)
Measure: Mean (Full Range); unit: years
Arm/Group | Randomized to GS First | Randomized to KS First
Number analyzed (Participants) | 7 | 6
years | 17 [4 to 29] | 17 [1 to 28]
Statistical Analysis 1: Comparison: Randomized to GS First vs Randomized to KS First; Test type: Superiority or Other; p > 0.05, Correlation — Correlation between years of experience (all anesthesiologists, pooled) and time to intubation (both GS and KS VLSs, pooled); R-squared = 0.16

6. Secondary Outcome: Number of Intubation Attempts to Reach "Best Obtainable Time to Intubation"
Description: For each anesthesiologist, the median time-to-intubation for patients #1-5, #6-10, #11-15, and #16-20 was determined. The anesthesiologist was considered to have reached "Best Obtainable Time (BOT) to Intubation" once the median time on any group of 5 consecutive patients was less than 3 seconds faster than the median time in the previous group of 5 consecutive patients, provided that there were no failed intubations or subsequent failed intubations using the same device.
Time Frame: less than 5 minutes per intubation
Measure: Number; unit: participants
Groups:
- GS Intubations: Anesthesiologists who intubated minimum 18 children with the GS VLS.
- KS Intubations: Anesthesiologists who intubated minimum 18 children with the KS VLS
Arm/Group | GS Intubations | KS Intubations
Number analyzed (Participants) | 10 | 11
participants
  BOT occurred on intubations #1-5 | 2 | 4
  BOT occurred on intubations #6-10 | 1 | 3
  BOT occurred on intubations #11-15 | 5 | 1
  BOT occurred on intubations #16-20 | 2 | 0
  BOT not yet achieved | 0 | 3

ADVERSE EVENTS:
Time Frame: Duration of intubation attempt (maximum 5 minutes)
Description: The incidence of trauma was recorded during the study. Failed intubation was one of the outcomes on the study so these events were not specifically recorded as adverse outcomes.
Arm/Group | Overall Anesthesiologists | Baseline Intubation Participants | KS Intubation Participants | GS Intubaton Participants
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/249 | 0/196 | 0/201
Other Adverse Events (participants affected / at risk) | 0/13 | 2/249 | 2/196 | 4/201
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Anesthesiologists (N=13) | Baseline Intubation Participants (N=249) | KS Intubation Participants (N=196) | GS Intubaton Participants (N=201)
Traumatic intubation (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2) | 4 (4) — Minor trauma was sustained on intubation attempts in two children at baseline, four with the GlideScope (GS) (on intubation attempts 5, 6, 8 and 18) and two with the Karl Storz Direct Coupled Interface(DCI)(KS) on intubation attempts 6 and 16).

LIMITATIONS AND CAVEATS:
Level of success could only be determined for the 8 anesthesiologists who completed minimum 18 intubations with the GS or KS video laryngoscope. Only 6 of 14 completed the whole study so had data could be used in comparing the two scopes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No